CLINICAL TRIAL: NCT03582098
Title: A Retrospective Observational Study to Evaluate the Clinical Outcomes and Routine Management of Patients With Chronic Lymphocytic Leukaemia Treated With Idelalisib and Rituximab in the United Kingdom (UK) and Ireland
Brief Title: Clinical Outcomes and Routine Management of Adults With Chronic Lymphocytic Leukaemia Treated With Idelalisib and Rituximab in the United Kingdom (UK) and Ireland
Acronym: RETRO-idel
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-UK-312-4639
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Chronic Lymphocytic Leukaemia
Keywords: Idelalisib; Zydelig
MeSH Terms: conditions — Leukemia, B-Cell | interventions — idelalisib; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idelalisib and Rituximab: Individuals who received treatment for CLL with at least one dose of idelalisib and rituximab in accordance with the marketing authorisation.
  Interventions: Drug: Idelalisib; Drug: Rituximab

INTERVENTIONS:
Drug: Idelalisib — Tablets were administered in accordance with the marketing authorization.
  Other Names: Zydelig®
Drug: Rituximab — Tablets were administered in accordance with the marketing authorization.

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of idelalisib and rituximab in adults with chronic lymphocytic leukaemia (CLL) in a real world setting

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL documented within medical records
* Individuals who have received treatment for CLL with at least one dose of idelalisib and rituximab in accordance with the marketing authorisation at the time of starting idelalisib treatment
* Idelalisib and rituximab initiated on or before 31 December 2017

Exclusion Criteria:

* Individuals who received idelalisib as part of an interventional clinical trial
* Individuals who received idelalisib for other indications including follicular lymphoma (FL)
* Individuals who previously received idelalisib in combination with ofatumumab
* Use of idelalisib which is not in accordance with its marketing authorisation at the time of starting idelalisib treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be identified by sites/hospitals as eligible for inclusion in the study by review of hospital records, including prescribing databases and by members of their direct care team and/or site personnel. The study will only include individuals who initiated idelalisib from September 2014, the date of marketing authorisation, up to and inclusive of 31 December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 3 months
  Overall Response Rate (ORR) is defined as the proportion of participants who achieve a clinical response as documented within their patient records after the initiation of treatment with idelalisib and rituximab during the observation period.

SECONDARY OUTCOMES:
Overall Survival | Up to 3 months
  Overall survival (OS) is defined as the interval from the initiation of idelalisib and rituximab to death from any cause
Progression-Free Survival | Up to 3 months
  Progression-free survival (PFS) is defined as the interval from the initiation of idelalisib and rituximab to the first documentation of definitive disease progression or death from any cause; definitive disease progression is CLL progression based on documentation in participant records
Time to Next Treatment | Up to 3 months
  Time to next treatment (TTNT) is defined as the interval from the initiation of treatment with idelalisib and rituximab to the initiation of next treatment
Duration of Response | Up to 3 months
  Duration of response (DOR) is defined as the interval from the first documentation of clinical response to the earlier of the first documentation of definitive disease progression or death from any cause
Overall Safety and Tolerability of Idelalisib and Rituximab as Measured by the Incidence of Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) | Up to 3 months
Starting Dose of Idelalisib | Up to 3 months
Proportion of Participants with Dose-Modifications, Treatment Interruptions and Discontinuations of Idelalisib | Up to 3 months
Proportion of Participants For Whom antibiotic Prophylactic Measures were Effective | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- St James Hospital, Dublin, Ireland
- United Kingdom (15):
  - NHS Grampian, Aberdeen
  - University Hospital of Wales, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - London Northwest University NHS Trust, Eastcote
  - Medway Maritime Hospital, Gillingham
  - Queen Alexandra Hospital, Harrow
  - King's College Hospital NHS Foundation Trust, London
  - Milton Keynes University Hospital, Milton Keynes
  - Oxford University Hospitals NHS Trust, Oxford
  - Whiston Hospital - St Helens And Knowsley Teaching Hospitals NHS Trust, Prescot
  - Southend University Hospital NHS Foundation Trust, Southend-on-Sea
  - Royal Marsden Hospital, Sutton
  - Singleton Hospital, Swansea
  - Royal Cornwall Hospital, Truro
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No